CLINICAL TRIAL: NCT03101267
Title: Phase 2 Dose-finding Study of ASP4070 - A Randomized, Double-blind, Placebo-controlled, Dose-finding Study in Patients With Cedar Pollinosis Using an Environmental Exposure Chamber -
Brief Title: A Dose-finding Study of ASP4070
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Immunomic Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4070-CL-0020
Record Dates: First submitted 2017-04-02; First posted 2017-04-05 (Actual); Results first posted 2020-06-30 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Cedar pollinosis; ASP4070; DNA plasmid vaccine
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ASP4070 4 mg (Experimental): Participants received ASP4070 4 mg 8 times by intradermal vaccination at 14-day intervals.
  Interventions: Drug: ASP4070
- ASP4070 1 mg (Experimental): Participants received ASP4070 1 mg 8 times by intradermal vaccination at 14-day intervals.
  Interventions: Drug: ASP4070
- Placebo (Placebo Comparator): Participants received Placebo 8 times by intradermal vaccination at 14-day intervals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP4070 — Intradermal vaccination at 2-week intervals
  Arms: ASP4070 1 mg; ASP4070 4 mg
Drug: Placebo — Intradermal vaccination at 2-week intervals
  Arms: Placebo

SUMMARY:
The objective of this study was to evaluate the efficacy, safety, and dose-response of ASP4070 vaccinated in patients with cedar pollinosis.

DETAILED DESCRIPTION:
Subjects were vaccinated with ASP4070 or placebo at 2 week intervals. Clinical symptoms were evaluated after cedar pollen exposure in a chamber at 4, 8 and 12 weeks after the last vaccination to identify the timing of the onset of therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has exhibited symptoms of cedar pollinosis, consisting of nasal symptoms (sneezing, nasal discharge or nasal obstruction) and eye symptoms (itchy eyes or watery eyes) during the pollen dispersal seasons in 2016 and 2017
* Subject who is positive for the Japanese red cedar (JRC) pollen-specific serum IgE antibody test
* At screening, subject whose score has worsened compared to baseline over 120 to 180 minutes after cedar pollen exposure in a chamber

Exclusion Criteria:

* Subject who has positive the test result of serum IgE antibody specific to other antigen than JRC pollen at screening
* Subject who has received specific immunotherapy (including desensitization therapy) for cedar pollinosis in the past
* Subject who has received specific or non-specific immunotherapy within 5 years prior to screening
* Subject who has received laser therapy or surgery for the treatment of nasal symptoms within 3 years prior to screening.
* Subject who has a history of allergic reactions such as anaphylactic shock and exanthema generalized caused by food and/or medical products in the past
* Subject who has a positive test result for hepatitis B surface (HBs) antigen or anti-hepatitis C virus (HCV) antibody
* Subject who has nasal disease that may interfere with the evaluation
* Subject who has autoimmune disease or other serious primary disease
* Subject who was diagnosed with immunodeficiency in the past
* Subject who has a complication of seasonal allergic rhinitis (due to allergens other than Japanese cedars or cypress), perennial allergic rhinitis, rhinitis medicamentosa, or non-allergic rhinitis that requires medical treatment
* Subject who has a complication of cardiovascular disease
* Subject who has a complication of hepatic disease
* Subject who has a complication of renal disease
* Subject who has a complication of respiratory disease
* Subject has a complication of malignant tumor or has been diagnosed with or has received treatment for malignant tumor within 5 years prior to the first vaccination of the study drug
* Subject who was diagnosed with schizophrenia, other mental conditions
* Subject who has a complication that may have an impact on the results of the local or systemic reaction
* Subject who has received a vaccination of Cry j 2-LAMP vaccine
* Subject who has participated in a clinical study of ASP4070 and received a vaccination of the study drug.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Shinjuku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 150 participants with cedar pollinosis were enrolled in this study. Participants were randomly allocated to 3 groups in a ratio of 1:1:1 to ASP4070 4 mg group, ASP4070 1 mg group or placebo group.
Pre-assignment Details: "Class of Japanese Red Cedar (JRC) pollen-specific Immunoglobulin E (IgE) antibody test at screening visit 1" and "Change from pre-exposure in mean total 3 nasal symptom (sneezing, nasal discharge and nasal congestion) score 120 to 180 minutes after start of cedar pollen exposure at screening visit 2" were used as stratification.
Period: Primary Study Period
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Started | 50 | 50 | 50
Completed | 47 | 48 | 47
Not Completed | 3 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 3
Not completed — Miscellaneous | 2 | 0 | 0
Period: Pollinosis Symptoms Survey Period
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Started | 47 | 48 | 47
Completed | 47 | 48 | 47
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) consisted of all participants who were vaccinated with the study drug at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: year] | 38.4 (8.6) | 38.1 (8.5) | 37.8 (9.3) | 38.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 26 | 90
  Male | 17 | 19 | 24 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 50 | 50 | 150
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 50 | 50 | 50 | 150
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Class of Japanese Red Cedar (JRC) Specific Immunoglobulin E (IgE) Antibody Test [Count of Participants; unit: Participants] — JRC specific IgE antibody test at screening visit 1 was showed. JRC specific IgE antibody was classified from Class 1 to Class 6. Participants with Class 1 and 2 was excluded in the enrollment. Population: Full Analysis Set (FAS) consisted of all participants who were randomized, were vaccinated with the study drug at least once, and had at least 1 measurement for efficacy evaluation obtained after vaccination of the study drug.
  Participants
    number analyzed (Participants) | 48 | 49 | 48 | 145
    3 | 26 | 26 | 26 | 78
    4 | 16 | 15 | 17 | 48
    5 | 3 | 6 | 4 | 13
    6 | 3 | 2 | 1 | 6
Change From Pre-exposure in Mean of Total 3 Nasal Symptom Score During 120 to 180 Minutes [Mean (Standard Deviation); unit: units on a scale] — At screening visit 2, participants were assessed for each symptom (sneezing, nasal discharge and nasal congestion) using the score from 0 (None; no symptoms) to 4 (Very severe) every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure. 3TNSS was a summed score of each symptom, and mean of 3TNSS at 120 to 180 min is the average of 5 timepoints of 3TNSS score, which ranged from 0 to 12. Higher 3TNSS score indicated greater disease activity. Population: FAS
  units on a scale
    number analyzed (Participants) | 48 | 49 | 48 | 145
    (all) | 4.79 (1.53) | 4.89 (1.31) | 4.78 (1.25) | 4.82 (1.36)

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-Exposure in Mean Total 3 Nasal Symptom Score (3TNSS) 120 to 180 Minutes After Start of Cedar Pollen Exposure on Day 183
Description: Participants were assessed for each symptom (sneezing, nasal discharge and nasal congestion) using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but does not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interferes with the activities of daily living).
  3TNSS was a summed score of each symptom, and mean of 3TNSS at 120 to 180 min is the average of 5 timepoints of 3TNSS score, which ranged from 0 to 12. Higher 3TNSS score indicated greater disease activity.
Time Frame: Day 183 at pre-exposure and 120 to 180 minutes after the start of cedar pollen exposure (5 samples 15 minutes apart)
Population: Full Analysis Set (FAS) consisted of all participants who were randomized, vaccinated with the study drug at least once, and had at least 1 measurement for efficacy evaluation obtained after vaccination of the study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale | 2.04 (1.30) | 1.91 (1.82) | 1.98 (1.34)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; 3TNSS treatment comparison; Test type: Superiority; p = 0.777, Mixed model for repeated measures (MMRM); The MMRM model included treatment group, stratification factors, analysis visit and interaction of treatment group and analysis visit; Adjusted mean difference = 0.09, 95% CI 2-sided [-0.52 to 0.69]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; 3TNSS treatment comparison; Test type: Superiority; p = 0.983, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.01, 95% CI [-0.61 to 0.59]

2. Secondary Outcome: Change From Pre-Exposure in Mean Total 4 Nasal Symptom Score (4TNSS) 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for each symptom (sneezing, nasal discharge, nasal congestion and itchy nose) using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living). 4TNSS was a summed score of each symptom, and mean of 4TNSS at 120 to 180 min is the average of 5 timepoints of 4TNSS score, which ranged from 0 to 16. Higher 4TNSS score indicated greater disease activity.
Time Frame: Pre-exposure and 120-180 minutes after the start of pollen exposure (5 samples 15 minutes apart) on Days 127, 155, and 183
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 4.21 (1.73) | 4.07 (2.69) | 4.02 (2.51)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 3.46 (2.09) | 3.20 (2.73) | 3.32 (2.00)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 2.71 (1.61) | 2.58 (2.50) | 2.62 (1.81)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; 4TNSS treatment comparison at day 127; Test type: Superiority; p = 0.710, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.17, 95% CI 2-sided [-0.75 to 1.10]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; 4TNSS treatment comparison at day 127; Test type: Superiority; p = 0.872, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.07, 95% CI 2-sided [-0.84 to 0.99]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; 4TNSS treatment comparison at day 155; Test type: Superiority; p = 0.701, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.18, 95% CI 2-sided [-0.73 to 1.08]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; 4TNSS treatment comparison at day 155; Test type: Superiority; p = 0.925, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.04, 95% CI [-0.95 to 0.86]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; 4TNSS treatment comparison at day 183; Test type: Superiority; p = 0.690, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.16, 95% CI 2-sided [-0.64 to 0.97]
Statistical Analysis 6: Comparison: ASP4070 4 mg vs Placebo; 4TNSS treatment comparison at day 183; Test type: Superiority; p = 0.868, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.07, 95% CI 2-sided [-0.73 to 0.87]

3. Secondary Outcome: Change From Pre-Exposure in Sneezing Score 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for sneezing using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure. The mean of score at 120 to 180 minutes was calculated.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living)
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 0.57 (0.57) | 0.47 (0.53) | 0.49 (0.52)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 0.46 (0.42) | 0.39 (0.37) | 0.39 (0.39)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 0.40 (0.41) | 0.28 (0.37) | 0.36 (0.32)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; Sneezing score treatment comparison at day 127; Test type: Superiority; p = 0.502, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.07, 95% CI 2-sided [-0.14 to 0.29]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; Sneezing score treatment comparison at day 127; Test type: Superiority; p = 0.879, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.02, 95% CI 2-sided [-0.23 to 0.20]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; Sneezing score treatment comparison at day 155; Test type: Superiority; p = 0.444, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.06, 95% CI 2-sided [-0.10 to 0.22]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; Sneezing score treatment comparison at day 155; Test type: Superiority; p = 0.987, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.00, 95% CI 2-sided [-0.16 to 0.16]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; Sneezing score treatment comparison at day 183; Test type: Superiority; p = 0.645, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.03, 95% CI 2-sided [-0.12 to 0.18]
Statistical Analysis 6: Comparison: ASP4070 1 mg vs Placebo; Sneezing score treatment comparison at day 183; Test type: Superiority; p = 0.357, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.07, 95% CI 2-sided [-0.22 to 0.08]

4. Secondary Outcome: Change From Pre-Exposure in Nasal Discharge Score 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for nasal discharge using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure. The mean of score at 120 to 180 minutes was calculated.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living)
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 1.54 (0.62) | 1.30 (0.93) | 1.42 (0.82)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 1.29 (0.69) | 1.12 (0.91) | 1.27 (0.80)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 0.96 (0.65) | 0.93 (0.86) | 0.87 (0.62)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; Nasal discharge score treatment comparison at day 127; Test type: Superiority; p = 0.472, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.12, 95% CI 2-sided [-0.20 to 0.44]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; Nasal discharge score treatment comparison at day 127; Test type: Superiority; p = 0.497, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.11, 95% CI 2-sided [-0.43 to 0.21]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; Nasal discharge score treatment comparison at day 155; Test type: Superiority; p = 0.821, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.04, 95% CI 2-sided [-0.28 to 0.36]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; Nasal discharge score treatment comparison at day 155; Test type: Superiority; p = 0.414, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.13, 95% CI 2-sided [-0.45 to 0.19]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; Nasal discharge score treatment comparison at day 183; Test type: Superiority; p = 0.414, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.12, 95% CI 2-sided [-0.17 to 0.41]
Statistical Analysis 6: Comparison: ASP4070 1 mg vs Placebo; Nasal discharge score treatment comparison at day 183; Test type: Superiority; p = 0.566, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.08, 95% CI 2-sided [-0.20 to 0.37]

5. Secondary Outcome: Change From Pre-Exposure in Mean Nasal Congestion Score 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for nasal congestion using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure. The mean of score at 120 to 180 minutes was calculated.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living)
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 1.14 (0.70) | 1.26 (0.89) | 1.18 (0.92)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 0.91 (0.68) | 0.90 (0.89) | 0.92 (0.77)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 0.68 (0.62) | 0.70 (0.78) | 0.75 (0.70)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; Nasal congestion score treatment comparison at day 127; Test type: Superiority; p = 0.822, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.04, 95% CI [-0.37 to 0.30]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; Nasal congestion score treatment comparison at day 127; Test type: Superiority; p = 0.587, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.09, 95% CI 2-sided [-0.24 to 0.42]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; Nasal congestion score treatment comparison at day 155; Test type: Superiority; p = 0.975, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.00, 95% CI 2-sided [-0.30 to 0.31]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; Nasal congestion score treatment comparison at day 155; Test type: Superiority; p = 0.980, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.00, 95% CI 2-sided [-0.31 to 0.31]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; Nasal congestion score treatment comparison at day 183; Test type: Superiority; p = 0.621, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.07, 95% CI 2-sided [-0.35 to 0.21]
Statistical Analysis 6: Comparison: ASP4070 1 mg vs Placebo; Nasal congestion score treatment comparison at day 183; Test type: Superiority; p = 0.831, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.03, 95% CI 2-sided [-0.31 to 0.25]

6. Secondary Outcome: Change From Pre-Exposure in Mean Itchy Nose Score 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for itchy nose using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure. The mean of score at 120 to 180 minutes was calculated.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living)
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 0.97 (0.64) | 1.03 (0.88) | 0.93 (0.89)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 0.80 (0.75) | 0.79 (0.91) | 0.74 (0.80)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 0.68 (0.56) | 0.67 (0.80) | 0.63 (0.66)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; Itchy nose score treatment comparison at day 127; Test type: Superiority; p = 0.864, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.03, 95% CI 2-sided [-0.29 to 0.35]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; Itchy nose score treatment comparison at day 127; Test type: Superiority; p = 0.502, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.11, 95% CI 2-sided [-0.21 to 0.43]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; Itchy nose score treatment comparison at day 155; Test type: Superiority; p = 0.652, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.07, 95% CI 2-sided [-0.25 to 0.40]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; Itchy nose score treatment comparison at day 155; Test type: Superiority; p = 0.633, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.08, 95% CI 2-sided [-0.25 to 0.41]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; Itchy nose score treatment comparison at day 183; Test type: Superiority; p = 0.596, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.07, 95% CI 2-sided [-0.20 to 0.35]
Statistical Analysis 6: Comparison: ASP4070 1 mg vs Placebo; Itchy nose score treatment comparison at day 183; Test type: Superiority; p = 0.621, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.07, 95% CI 2-sided [-0.21 to 0.34]

7. Secondary Outcome: Change From Pre-Exposure in Mean Total Non-Nasal Symptom Score (TNNSS) 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for each non-nasal symptom (itchy eyes and watery eyes) using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living).
  TNNSS was a summed score of each symptom, and mean of TNNSS at 120 to 180 min is the average of 5 timepoints of TNNSS score, which ranged from 0 to 8. Higher TNNSS score indicated greater disease activity.
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 0.83 (1.22) | 0.96 (1.17) | 0.61 (0.93)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 0.62 (1.10) | 0.83 (1.40) | 0.50 (0.71)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 0.59 (1.09) | 0.73 (1.19) | 0.40 (0.71)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; TNNSS treatment comparison at day 127; Test type: Superiority; p = 0.336, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.21, 95% CI 2-sided [-0.22 to 0.65]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; TNNSS treatment comparison at day 127; Test type: Superiority; p = 0.102, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.36, 95% CI 2-sided [-0.07 to 0.80]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; TNNSS treatment comparison at day 155; Test type: Superiority; p = 0.625, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.11, 95% CI 2-sided [-0.34 to 0.56]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; TNNSS treatment comparison at day 155; Test type: Superiority; p = 0.145, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.33, 95% CI 2-sided [-0.12 to 0.78]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; TNNSS treatment comparison at day 183; Test type: Superiority; p = 0.364, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.19, 95% CI 2-sided [-0.22 to 0.59]
Statistical Analysis 6: Comparison: ASP4070 1 mg vs Placebo; TNNSS treatment comparison at day 183; Test type: Superiority; p = 0.082, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.35, 95% CI 2-sided [-0.05 to 0.76]

8. Secondary Outcome: Change From Pre-Exposure in Mean Itchy Eyes Score 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for itchy eyes using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure. The mean of score at 120 to 180 minutes was calculated.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living)
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 0.51 (0.75) | 0.58 (0.72) | 0.44 (0.66)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 0.36 (0.63) | 0.49 (0.80) | 0.33 (0.50)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 0.35 (0.67) | 0.43 (0.69) | 0.29 (0.51)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; Itchy eyes treatment comparison at day 127; Test type: Superiority; p = 0.623, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.07, 95% CI 2-sided [-0.21 to 0.35]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; Itchy eyes treatment comparison at day 127; Test type: Superiority; p = 0.288, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.15, 95% CI 2-sided [-0.13 to 0.43]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; Itchy eyes treatment comparison at day 155; Test type: Superiority; p = 0.830, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.03, 95% CI 2-sided [-0.24 to 0.30]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; Itchy eyes treatment comparison at day 155; Test type: Superiority; p = 0.208, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.17, 95% CI 2-sided [-0.10 to 0.44]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; Itchy eyes treatment comparison at day 183; Test type: Superiority; p = 0.616, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.06, 95% CI 2-sided [-0.19 to 0.31]
Statistical Analysis 6: Comparison: ASP4070 1 mg vs Placebo; Itchy eyes treatment comparison at day 183; Test type: Superiority; p = 0.207, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.16, 95% CI 2-sided [-0.09 to 0.41]

9. Secondary Outcome: Change From Pre-Exposure in Mean Watery Eyes Score 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for watery eyes using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure. The mean of score at 120 to 180 minutes was calculated.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living)
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 0.32 (0.57) | 0.38 (0.57) | 0.17 (0.38)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 0.26 (0.55) | 0.34 (0.67) | 0.17 (0.37)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 0.24 (0.48) | 0.30 (0.57) | 0.11 (0.29)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; Watery eyes treatment comparison at day 127; Test type: Superiority; p = 0.157, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.15, 95% CI 2-sided [-0.06 to 0.35]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; Watery eyes treatment comparison at day 127; Test type: Superiority; p = 0.039, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.21, 95% CI 2-sided [0.01 to 0.41]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; Watery eyes treatment comparison at day 155; Test type: Superiority; p = 0.459, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.08, 95% CI 2-sided [-0.14 to 0.30]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; Watery eyes treatment comparison at day 155; Test type: Superiority; p = 0.153, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.16, 95% CI 2-sided [-0.06 to 0.38]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; Watery eyes treatment comparison at day 183; Test type: Superiority; p = 0.195, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.12, 95% CI 2-sided [-0.06 to 0.31]
Statistical Analysis 6: Comparison: ASP4070 1 mg vs Placebo; Watery eyes treatment comparison at day 183; Test type: Superiority; p = 0.038, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.20, 95% CI 2-sided [0.01 to 0.38]

10. Secondary Outcome: Change From Pre-Exposure in Total 5 Symptom Score (5TSS) 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for each 5TSS (sneezing, nasal discharge, nasal congestion, itchy eyes and watery eyes) using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living).
  5TSS was a summed score of each symptom, and mean of 5TSS at 120 to 180 min is the average of 5 timepoints of 5TSS score, which ranged from 0 to 20. Higher 5TSS score indicated greater disease activity.
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 4.08 (1.95) | 3.99 (2.67) | 3.70 (2.40)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 3.28 (2.07) | 3.24 (2.98) | 3.07 (1.84)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 2.63 (1.82) | 2.64 (2.62) | 2.38 (1.68)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; 5TSS treatment comparison at day 127; Test type: Superiority; p = 0.433, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.37, 95% CI 2-sided [-0.56 to 1.29]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; 5TSS treatment comparison at day 127; Test type: Superiority; p = 0.479, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.33, 95% CI 2-sided [-0.59 to 1.24]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; 5TSS treatment comparison at day 155; Test type: Superiority; p = 0.648, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.22, 95% CI 2-sided [-0.71 to 1.14]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; 5TSS treatment comparison at day 155; Test type: Superiority; p = 0.654, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.21, 95% CI 2-sided [-0.72 to 1.14]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; 5TSS treatment comparison at day 183; Test type: Superiority; p = 0.514, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.27, 95% CI 2-sided [-0.55 to 1.09]
Statistical Analysis 6: Comparison: ASP4070 1 mg vs Placebo; 5TSS treatment comparison at day 183; Test type: Superiority; p = 0.400, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.35, 95% CI 2-sided [-0.47 to 1.17]

11. Secondary Outcome: Change From Pre-Exposure in Mean Total 6 Symptom Score (6TSS) 120 to 180 Minutes After Cedar Pollen Exposure
Description: Participants were assessed for each 6TSS (sneezing, nasal discharge, nasal congestion, itchy nose, itchy eyes and watery eyes) using the following score every 15 minutes from before cedar pollen exposure until 180 minutes after cedar pollen exposure.
  0: None (no symptoms)
  1. Mild (symptoms present but easily tolerated)
  2. Moderate (awareness of symptoms; bothersome, but tolerable)
  3. Severe (definite awareness of symptoms; difficult to tolerate, but did not interfere with the activities of daily living)
  4. Very severe (difficult to tolerate and interfered with the activities of daily living).
  6TSS was a summed score of each symptom, and mean of 6TSS at 120 to 180 min is the average of 5 timepoints of 6TSS score, which ranged from 0 to 24. Higher 6TSS score indicated greater disease activity.
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Day 127: number analyzed (Participants) | 47 | 49 | 48
  Day 127 | 5.04 (2.39) | 5.02 (3.31) | 4.63 (3.09)
  Day 155: number analyzed (Participants) | 47 | 47 | 46
  Day 155 | 4.08 (2.66) | 4.03 (3.74) | 3.82 (2.30)
  Day 183: number analyzed (Participants) | 47 | 48 | 47
  Day 183 | 3.30 (2.19) | 3.31 (3.29) | 3.02 (2.14)
Statistical Analysis 1: Comparison: ASP4070 4 mg vs Placebo; 6TSS treatment comparison at day 127; Test type: Superiority; p = 0.505, MMRM — The MMRM model included treatment group, stratification factors, analysis visit and interaction of treatment group and analysis visit; Adjusted mean difference, = 0.39, 95% CI 2-sided [-0.76 to 1.54]
Statistical Analysis 2: Comparison: ASP4070 1 mg vs Placebo; 6TSS treatment comparison at day 127; Test type: Superiority; p = 0.451, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference, = 0.44, 95% CI 2-sided [-0.71 to 1.58]
Statistical Analysis 3: Comparison: ASP4070 4 mg vs Placebo; 6TSS treatment comparison at day 155; Test type: Superiority; p = 0.623, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference, = 0.29, 95% CI 2-sided [-0.88 to 1.46]
Statistical Analysis 4: Comparison: ASP4070 1 mg vs Placebo; 6TSS treatment comparison at day 155; Test type: Superiority; p = 0.620, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference, = 0.29, 95% CI 2-sided [-0.87 to 1.46]
Statistical Analysis 5: Comparison: ASP4070 4 mg vs Placebo; 6TSS treatment comparison at day 183; Test type: Superiority; p = 0.504, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference, = 0.35, 95% CI 2-sided [-0.68 to 1.37]
Statistical Analysis 6: Comparison: ASP4070 1 mg vs Placebo; 6TSS treatment comparison at day 183; Test type: Superiority; p = 0.414, MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference, = 0.42, 95% CI 2-sided [-0.60 to 1.45]

12. Secondary Outcome: Time to Occurrence of Nasal or Eye Symptom From Start of Cedar Pollen Exposure
Description: Time point when the score of nasal or eye symptom worsens by 1 or more as compared to before cedar pollen exposure were assessed.
Time Frame: Days 127, 155 and 183, from the start of cedar pollen exposure for up to 180 minutes
Population: FAS
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
minutes
  Day 127: number analyzed (Participants) | 47 | 48 | 48
  Day 127 | 15.0 [15.0 to 30.0] | 15.0 [15.0 to 30.0] | 30.0 [15.0 to 30.0]
  Day 155: number analyzed (Participants) | 48 | 44 | 45
  Day 155 | 22.5 [15.0 to 30.0] | 30.0 [15.0 to 30.0] | 15.0 [15.0 to 30.0]
  Day 183: number analyzed (Participants) | 47 | 43 | 44
  Day 183 | 30.0 [NA to NA] — 95% Confidential Interval (CI) was not technically defined due to insufficient number of participants with events around the percentile. | 30.0 [15.0 to 45.0] | 30.0 [NA to NA] — 95% Confidential Interval (CI) was not technically defined due to insufficient number of participants with events around the percentile.

13. Secondary Outcome: Amount of Nasal Discharge Per 30 Minutes During Cedar Pollen Exposure
Description: Nasal discharge amount was calculated by the difference in the weight of the tissue paper before and after use by participants who were instructed to use pre-allocated tissues for blowing their nose.
Time Frame: Day 127: 0-30 min, 30-60 min, 60-90 min, 90-120 min, 120-150 min, 150-180 min, Day 155: 0-30 min, 30-60 min, 60-90 min, 90-120 min, 120-150 min, 150-180 min, Day 183: 0-30 min, 30-60 min, 60-90 min, 90-120 min, 120-150 min, 150-180 min
Population: FAS
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
gram
  Day 127: 0-30 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 0-30 min | 0.57 (0.90) | 0.80 (1.31) | 0.68 (1.11)
  Day 127: 30-60 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 30-60 min | 1.21 (1.06) | 1.35 (1.74) | 1.43 (1.58)
  Day 127: 60-90 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 60-90 min | 1.58 (1.41) | 1.61 (1.91) | 1.73 (1.88)
  Day 127: 90-120 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 90-120 min | 1.72 (1.53) | 1.43 (1.76) | 1.67 (2.24)
  Day 127: 120-150 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 120-150 min | 1.49 (1.28) | 1.59 (1.96) | 1.67 (1.89)
  Day 127: 150-180 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 150-180 min | 1.64 (1.42) | 1.56 (1.77) | 1.61 (1.79)
  Day 155: 0-30 min: number analyzed (Participants) | 48 | 47 | 46
  Day 155: 0-30 min | 0.55 (1.88) | 0.79 (1.66) | 0.91 (1.52)
  Day 155: 30-60 min: number analyzed (Participants) | 48 | 47 | 46
  Day 155: 30-60 min | 1.12 (1.31) | 1.23 (1.72) | 1.57 (1.64)
  Day 155: 60-90 min: number analyzed (Participants) | 48 | 47 | 46
  Day 155: 60-90 min | 1.25 (1.46) | 1.45 (2.08) | 1.75 (1.84)
  Day 155: 90-120 min: number analyzed (Participants) | 48 | 47 | 46
  Day 155: 90-120 min | 1.42 (1.79) | 1.62 (2.24) | 1.71 (1.89)
  Day 155: 120-150 min: number analyzed (Participants) | 47 | 47 | 46
  Day 155: 120-150 min | 1.45 (1.57) | 1.82 (2.59) | 1.83 (2.00)
  Day 155: 150-180 min: number analyzed (Participants) | 47 | 47 | 46
  Day 155: 150-180 min | 1.63 (1.69) | 1.91 (2.56) | 1.70 (2.00)
  Day 183: 0-30 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 0-30 min | 0.35 (0.92) | 0.44 (0.89) | 0.49 (1.16)
  Day 183: 30-60 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 30-60 min | 0.57 (1.00) | 0.73 (1.08) | 0.90 (1.39)
  Day 183: 60-90 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 60-90 min | 0.71 (0.94) | 1.20 (1.93) | 0.84 (0.98)
  Day 183: 90-120 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 90-120 min | 0.94 (1.23) | 1.23 (2.02) | 0.90 (1.02)
  Day 183: 120-150 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 120-150 min | 1.13 (1.52) | 1.42 (2.18) | 1.05 (1.18)
  Day 183: 150-180 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 150-180 min | 1.06 (1.35) | 1.54 (2.07) | 1.23 (1.34)

14. Secondary Outcome: Sneezing Count Per 30 Minutes During Cedar Pollen Exposure
Description: Sneezing count per 30 minutes were measured during chamber exposure.
Time Frame: as for outcome 13
Population: FAS
Measure: Mean (Standard Deviation); unit: sneezes
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48
sneezes
  Day 127: 0-30 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 0-30 min | 0.4 (0.7) | 0.8 (0.9) | 1.1 (2.1)
  Day 127: 30-60 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 30-60 min | 1.0 (1.2) | 1.0 (1.5) | 1.3 (2.8)
  Day 127: 60-90 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 60-90 min | 1.4 (2.0) | 1.5 (2.0) | 1.3 (1.6)
  Day 127: 90-120 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 90-120 min | 1.4 (1.9) | 1.2 (2.4) | 1.7 (2.5)
  Day 127: 120-150 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 120-150 min | 1.5 (2.6) | 1.4 (2.1) | 1.3 (2.2)
  Day 127: 150-180 min: number analyzed (Participants) | 47 | 49 | 48
  Day 127: 150-180 min | 1.6 (2.1) | 1.2 (1.7) | 1.5 (2.1)
  Day 155: 0-30 min: number analyzed (Participants) | 48 | 47 | 46
  Day 155: 0-30 min | 0.8 (1.1) | 0.6 (0.8) | 0.8 (1.4)
  Day 155: 30-60 min: number analyzed (Participants) | 48 | 47 | 46
  Day 155: 30-60 min | 0.9 (1.2) | 1.0 (1.4) | 1.1 (2.5)
  Day 155: 60-90 min: number analyzed (Participants) | 48 | 47 | 46
  Day 155: 60-90 min | 1.0 (1.1) | 1.1 (1.4) | 1.1 (1.6)
  Day 155: 90-120 min: number analyzed (Participants) | 47 | 47 | 46
  Day 155: 90-120 min | 1.0 (1.8) | 1.1 (1.9) | 1.0 (1.3)
  Day 155: 120-150 min: number analyzed (Participants) | 47 | 47 | 46
  Day 155: 120-150 min | 1.1 (1.3) | 1.0 (1.3) | 1.3 (1.5)
  Day 155: 150-180 min: number analyzed (Participants) | 47 | 47 | 46
  Day 155: 150-180 min | 1.4 (2.0) | 1.0 (1.4) | 1.0 (1.7)
  Day 183: 0-30 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 0-30 min | 0.6 (1.0) | 0.6 (1.0) | 0.5 (0.8)
  Day 183: 30-60 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 30-60 min | 0.7 (1.3) | 0.4 (0.8) | 0.6 (0.9)
  Day 183: 60-90 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 60-90 min | 0.8 (0.9) | 0.7 (1.0) | 0.9 (1.5)
  Day 183: 90-120 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 90-120 min | 1.0 (1.3) | 0.7 (1.1) | 0.9 (1.3)
  Day 183: 120-150 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 120-150 min | 1.1 (1.5) | 0.7 (1.0) | 1.1 (1.5)
  Day 183: 150-180 min: number analyzed (Participants) | 47 | 48 | 47
  Day 183: 150-180 min | 0.9 (1.4) | 0.8 (1.3) | 1.0 (1.2)

15. Secondary Outcome: Number of Participants With Adverse Events (AE) During the Primary Study Period
Description: Treatment emergent adverse events (TEAE) was defined as an AE observed after starting administration of the test drug/comparative drug. A drug-related TEAE was a TEAE with either possible or probable relationship to the study drug as assessed by the investigator. Severity of AEs was assessed according to the following 4 levels. Mild: no disruption of normal daily activities, Moderate: affect normal daily activities, Severe: inability to perform daily activities, Life-threatening: necessity for urgent intervention.
  If the investigator or subinvestigator examined the patient and determined that the following items occurred from the date of study drug vaccination until 14 days after vaccination and a relationship with the study drug could not be negated, then it was evaluated as a local/systemic reaction at the vaccination site.
  * Local reactions: pain, tenderness, erythema/redness and induration/swelling
  * Systemic reactions: nausea/vomiting, diarrhea, headache, fatigue and myalgia
Time Frame: From first dose of study drug up to the end of primary study period (up to 7 days after Day 183)
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 50 | 50 | 50
Participants
  TEAE | 49 | 44 | 28
  Mild | 33 | 33 | 18
  Moderate | 13 | 11 | 10
  Severe | 3 | 0 | 0
  Life-threatening Possibility | 0 | 0 | 0
  Drug-related TEAE | 45 | 37 | 18
  Device-Related TEAE | 0 | 0 | 0
  Serious TEAE | 2 | 0 | 0
  Drug-related serious TEAE | 0 | 0 | 0
  TEAE leading to withdrawal of treatment | 0 | 0 | 0
  Drug-related TEAE leading to withdrawal of treat. | 0 | 0 | 0
  Death | 0 | 0 | 0
  Local reaction | 34 | 24 | 7
  Systemic reaction | 13 | 13 | 9
  TEAEs other than local or systemic reactions | 48 | 40 | 21
  Drug-related TEAEs other than local or systemic | 38 | 31 | 6

16. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE) During the Long-Term Safety Follow-Up Period
Description: If SAEs occurred, then the participant was to contact the study site. With regard to participants who had discontinued the study during the primary study period, if the study drug had been vaccinated even once, then safety information (SAEs) was collected for 1 year after the final vaccination.
Time Frame: Up to 9 months after the end of primary study period (primary study period was up to 7 days after Day 183)
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
Number analyzed (Participants) | 50 | 50 | 50
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to the end of primary study period (up to 7 days after Day 183). SAEs were collected up to 9 months after the end of primary study period (until 12 months after the final vaccination of the study drug).
Description: SAF consisted of all participants who were vaccinated with the study drug at least once.
Arm/Group | ASP4070 4 mg | ASP4070 1 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 47/50 | 41/50 | 23/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP4070 4 mg (N=50) | ASP4070 1 mg (N=50) | Placebo (N=50)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP4070 4 mg (N=50) | ASP4070 1 mg (N=50) | Placebo (N=50)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Fatigue (General disorders) | 5 (13) | 6 (19) | 7 (8)
Induration (General disorders) | 8 (24) | 2 (6) | 0 (0)
Pain (General disorders) | 11 (32) | 5 (10) | 1 (1)
Swelling (General disorders) | 8 (14) | 1 (2) | 0 (0)
Tenderness (General disorders) | 23 (71) | 13 (62) | 5 (6)
Vaccination site pruritus (General disorders) | 37 (179) | 29 (134) | 0 (0)
Nasopharyngitis (Infections and infestations) | 18 (19) | 11 (12) | 9 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 8 (13) | 14 (27) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 31 (146) | 15 (43) | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT03101267/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03101267/SAP_001.pdf